CLINICAL TRIAL: NCT01918982
Title: Interest of Circulating Endothelial Progenitor Cells CD34+144+CD14- and CD34+VEGF-R2+CD14- in the Follow-up of Aortic Aneurysm
Brief Title: Circulating Endothelial Progenitor Cells and Aortic Aneurysm
Acronym: ANOPEC3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hopital Jean Minjoz (Other)
Responsible Party: Principal Investigator, Prof. Sidney Chocron, MD, PhD, Hopital Jean Minjoz
Other Study IDs: 147/362
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: - Aortic Aneurysm
Keywords: Aortic aneurysm; circulating endothelial progenitor cells
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic aneurysm: Patients with aortic aneurysm >30mm and < 50mm

SUMMARY:
We aimed to see if aortic aneurysms could be followed-up by circulating endothelial progenitor cells CD34+144+CD14- and CD34+VEGF-R2+CD14- blood level.

DETAILED DESCRIPTION:
Circulating endothelial progenitor cells CD34+144+CD14- and CD34+VEGF-R2+CD14- have been shown to be inversely correlated to aortic aneurysm size. We aimed to see if aortic aneurysms could be followed-up by circulating endothelial progenitor cells CD34+144+CD14- and CD34+VEGF-R2+CD14- blood level. 40 patients followed for known aortic aneurysm >30mm and <50mm will be followed up every 6 months during 2 years. Each 6 months they will have a consultation by their physiologist with an echo or a CT-scan. At the same time, a 10ML blood sample will be taken to assess the circulating endothelial progenitor cells CD34+144+CD14- and CD34+VEGF-R2+CD14- blood level.

ELIGIBILITY:
Inclusion Criteria:

* Aortic aneurysm size >30mm and > 50mm

Exclusion Criteria:

* Infectious disease
* Inflammatory disease
* Liver insuffisency
* Cancer evolutive
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Circulating endothelial progenitor cells CD34+144+CD14- and CD34+VEGF-R2+CD14- blood concentration | 2 years
  Patients are followed for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Chocron, MD, PhD, Principal Investigator — Université de Franche-comté. France; Andrea Perrotti, MD, Principal Investigator — Université de Franche-Comté. France; Simon Rinckenbach, MD, PhD, Principal Investigator — Université de Franche-Comté. France; Siamak Davani, MD, PhD, Principal Investigator — Université de Franche-Comté. France

REFERENCES:
- [Background] Parietti E, Pallandre JR, Deschaseaux F, Aupecle B, Durst C, Kantelip JP, Chocron S, Davani S. Presence of circulating endothelial progenitor cells and levels of stromal-derived factor-1alpha are associated with ascending aorta aneurysm size. Eur J Cardiothorac Surg. 2011 Jul;40(1):e6-12. doi: 10.1016/j.ejcts.2011.02.065. Epub 2011 Apr 9. PMID 21481600